CLINICAL TRIAL: NCT03174613
Title: A Dose Blocked-randomized, Double-blind, Placebo Controlled, Single and Multiple Dosing, Dose-escalation Phase I Clinical Trial to Investigate the Safety, Tolerability, Pharmacokinetic/Pharmacodynamics and Food Effect of LC51-0255
Brief Title: A Study To Evaluate The Safety, Pharmacokinetics/Pharmacodynamics (PK/PD) and Food Effect Of LC51-0255
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: LG Chem (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: LG-SGCL001
Record Dates: First submitted 2017-05-25; First posted 2017-06-02 (Actual); Last update posted 2020-09-18 (Actual); Status verified 2020-09

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Double blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- LC51-0255 (Experimental): tablets, PO
  Interventions: Drug: LC51-0255
- Placebo (Placebo Comparator): tablets, PO
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: LC51-0255 — 0.25mg, 0.5mg, 1mg, 2mg, 4mg, 8mg
  Arms: LC51-0255
Drug: Placebo — 0.25mg, 0.5mg, 1mg, 2mg, 4mg, 8mg
  Arms: Placebo

SUMMARY:
1. To evaluate the safety and tolerability of LC51-0255 in healthy male subjects
2. To evaluate the pharmacokinetic/pharmacodynamics characteristics (PK/PD) of LC51-0255 in healthy male subjects
3. To evaluate bioavailability of LC51-0255

DETAILED DESCRIPTION:
For safety and tolerability assessement, subjects will be monitored by collection of adverse events, physical exams, vital sign, 12-Lead ECG, Continuous ECG monitoring, Holter monitoring, blood chemistry and hematology panels, pulmonary function tests, optical coherence tomography (OCT) during the study.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male subjects aged 19~45 years at screening.
* Subjects with BMI between 18.0(inclusive) and 27.0 kg/m2 (exclusive)

Exclusion Criteria:

* History or Known presence of clinically relevant hepatic, gastrointestinal, pulmonary, psychiatric, endocrine, neurological, cancer, including solid tumors and hematological malignancies, cardiovascular, ophthalmological or other major systemic disease
* Exclusions Related to Laboratory Results: Platelet count < 100,000/μL, Hgb < 8.5 g/dL, Neutrophils < 1.5 /μL, Absolute WBC count < 3500/μL, Absolute lymphocyte count < 800/μL

Ages: 19 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Healthy male subjects
Enrollment: 100 (Actual)
Dates: Start 2017-05-31 (Actual); Primary Completion 2019-06-12 (Actual); Study Completion 2019-07-11 (Actual)

PRIMARY OUTCOMES:
MTD determination | Dose limiting Toxicity will be evaluated at Day 19 in Single dosing study and at Day 39 in Multiple dosing study
  Safety and Tolerability

SECONDARY OUTCOMES:
Pharmacokinetic: Peak Plasma Concentration (Cmax) | Cmax:168 hours post dose
  Cmax
Pharmacokinetic: Area under the plasma concentration versus time curve (AUC) | AUCinf:168 hours post dose
  AUC

CONTACTS AND LOCATIONS:
Overall Officials: Kyung-Sang Yu, MD,M.B.A., Principal Investigator — Seoul National University Hospital, Clinical Trial Center
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No